CLINICAL TRIAL: NCT00372385
Title: A Phase 2 Study of VX-950 in Combination With Peginterferon Alfa-2a (Pegasys®), With and Without Ribavirin (Copegus®) in Subjects With Hepatitis C
Brief Title: Phase 2 Study of VX-950, Pegasys® With and Without Copegus® in Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX05-950-104EU
Record Dates: First submitted 2006-09-01; First posted 2006-09-06 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; telaprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (Placebo Comparator): Placebo (PBO) matched to telaprevir tablet orally thrice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 48 weeks.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a; Drug: Placebo
- Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet orally thrice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 weeks.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a; Drug: Telaprevir
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 12 weeks.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a; Drug: Telaprevir
- Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection, for 12 weeks.
  Interventions: Drug: Pegylated Interferon Alfa 2a; Drug: Telaprevir

INTERVENTIONS:
Drug: Ribavirin — tablet
  Arms: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week; Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Drug: Pegylated Interferon Alfa 2a — Solution for injection
Drug: Placebo — tablet
  Arms: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week
Drug: Telaprevir — tablet
  Other Names: VX-950
  Arms: Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week

SUMMARY:
Compare the effectiveness of telaprevir (VX-950) in combination with Pegylated Interferon Alfa 2a (Peg-IFN-alfa-2a) with and without Ribavirin (RBV) in reducing plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus Genotype 1 with detectable plasma hepatitis C virus RNA
* Have been infected with Hepatitis C virus for greater than (>) 6 months
* Seronegative for hepatitis B surface antigen and human immunodeficiency virus 1 and 2
* Must agree to use 2 methods of contraception, including 1 barrier method, during and for 24 weeks after the completion of the study (unless the subject is a female of documented non-child-bearing potential)
* Female subjects must have a negative pregnancy test at all visits before the first dose.

Exclusion Criteria:

* Received any approved or investigational drug or drug regimen for the treatment of hepatitis C.
* Any medical contraindications to Peg-IFN-alfa-2a or Ribavirin therapy
* Any other cause of significant liver disease in addition to hepatitis C; this may include but is not limited to, hepatitis B, drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, Nonalcoholic Steatohepatitis or primary biliary cirrhosis.
* Diagnosed or suspected hepatocellular carcinoma.
* Histologic evidence of hepatic cirrhosis (including compensated cirrhosis) based on a liver biopsy taken within 2 years before Study start.
* Alcohol/drug abuse or excessive use in the last 12 months.
* Participation in any investigational drug study within 90 days before drug administration or participation in more than 2 drug studies in the last 12 months (exclusive of the current study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (4):
- Call For Information, Call For Information, Austria
- Call For Information, Call For Information, France
- Call For Information, Call For Information, Germany
- Call for Information, Call For Information, United Kingdom

REFERENCES:
- [Derived] Hezode C, Forestier N, Dusheiko G, Ferenci P, Pol S, Goeser T, Bronowicki JP, Bourliere M, Gharakhanian S, Bengtsson L, McNair L, George S, Kieffer T, Kwong A, Kauffman RS, Alam J, Pawlotsky JM, Zeuzem S; PROVE2 Study Team. Telaprevir and peginterferon with or without ribavirin for chronic HCV infection. N Engl J Med. 2009 Apr 30;360(18):1839-50. doi: 10.1056/NEJMoa0807650. PMID 19403903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 334 subjects were enrolled, of which 11 subjects discontinued the study prior to study drug administration. A total of 323 subjects started treatment.
Period: Overall Study
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Started | 82 | 81 | 82 | 78
Completed | 49 | 61 | 72 | 70
Not Completed | 33 | 20 | 10 | 8
Not completed — Adverse Event | 6 | 11 | 9 | 7
Not completed — Noncompliance | 0 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Refusal of Treatment | 3 | 6 | 0 | 0
Not completed — No Response | 1 | 1 | 0 | 0
Not completed — Ineligibility due to Exclusion Criterion | 1 | 0 | 0 | 0
Not completed — Virologic Stopping Rule | 17 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week | Total
Number analyzed (Participants) | 82 | 81 | 82 | 78 | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 81 | 80 | 81 | 78 | 320
  >=65 years | 0 | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.6) | 44.3 (10.0) | 44.1 (10.2) | 44.3 (10.8) | 44.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 27 | 33 | 35 | 131
  Male | 46 | 54 | 49 | 43 | 192
Region of Enrollment [Number; unit: participants]
  Europe | 82 | 81 | 82 | 78 | 323

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 24 After the Completion of Study Drug Dosing
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: 24 weeks after the completion of study drug dosing (up to Week 72)
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Number analyzed (Participants) | 82 | 81 | 82 | 78
percentage of participants | 46.3 [35 to 58] | 69.1 [58 to 79] | 59.8 [48 to 70] | 35.9 [25 to 48]
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Test type: Superiority or Other; p = 0.0026, Regression, Logistic; Odds Ratio (OR) = 2.758, 95% CI 2-sided [1.424 to 5.340]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week; Test type: Superiority or Other; p = 0.959, Regression, Logistic; Odds Ratio (OR) = 1.709, 95% CI 2-sided [0.910 to 3.212]
Statistical Analysis 3: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week; Test type: Superiority or Other; p = 0.1089, Regression, Logistic; Odds Ratio (OR) = 0.589, 95% CI 2-sided [0.309 to 1.125]

2. Secondary Outcome: Percentage of Subjects With Undetectable Plasma HCV RNA at Week 12 After the Completion of Study Drug Dosing
Description: as for outcome 1
Time Frame: 12 weeks after the completion of study drug dosing (up to Week 60)
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Number analyzed (Participants) | 82 | 81 | 82 | 78
percentage of participants | 47.6 [36 to 59] | 69.1 [58 to 79] | 59.8 [48 to 70] | 37.2 [26 to 49]
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Test type: Superiority or Other; p = 0.0041, Regression, Logistic; Odds Ratio (OR) = 2.632, 95% CI 2-sided [1.359 to 5.097]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week; Test type: Superiority or Other; p = 0.1324, Regression, Logistic; Odds Ratio (OR) = 1.623, 95% CI 2-sided [0.864 to 3.050]
Statistical Analysis 3: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week; Test type: Superiority or Other; p = 0.1099, Regression, Logistic; Odds Ratio (OR) = 0.591, 95% CI 2-sided [0.311 to 1.126]

3. Secondary Outcome: Percentage of Subjects With Undetectable Plasma HCV RNA at Completion of Study Drug Dosing
Description: as for outcome 1
Time Frame: Completion of study drug dosing (up to Week 48)
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Number analyzed (Participants) | 82 | 81 | 82 | 78
percentage of participants | 54.9 [43 to 66] | 70.4 [59 to 80] | 80.5 [70 to 88] | 61.5 [50 to 72]

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline up to Week 48
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Number analyzed (Participants) | 82 | 81 | 82 | 78
participants
  AEs | 81 | 80 | 82 | 78
  SAEs | 8 | 16 | 11 | 9

5. Secondary Outcome: Number of Subjects With Viral Relapse
Description: Viral relapse was defined as having detectable HCV RNA during antiviral follow-up. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: After last dose of study drug up to antiviral follow-up (up to Week 72)
Population: Analysis population included subjects who completed their assigned study drug treatment and had undetectable HCV RNA at the completion of treatment (up to Week 48).
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Number analyzed (Participants) | 45 | 57 | 63 | 46
participants | 10 | 8 | 19 | 22

6. Secondary Outcome: Maximum (Cmax), Minimum (Cmin) and Average (Cavg) Plasma Concentration of Telaprevir
Description: Only subjects who received telaprevir were to be analyzed for this outcome. Maximum, minimum and average plasma concentrations observed during assessment period were reported.
Time Frame: Day 1, 4, 8, 15, 22, 29, 43, 57, 71, 85
Population: Pharmacokinetic population included all subjects who provided pharmacokinetic assessments and had evaluable and interpretable data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Telaprevir: All Subjects from "Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week" and "Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week" reporting groups who received single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks.
Arm/Group | Telaprevir
Number analyzed (Participants) | 239
nanogram per milliliter (ng/mL)
  Cmax | 3370 (755)
  Cmin | 2510 (604)
  Cavg | 3055 (694)

ADVERSE EVENTS:
Time Frame: Adverse Events during Baseline through Week 48
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week
Serious Adverse Events (participants affected / at risk) | 8/82 | 16/81 | 11/82 | 9/78
Other Adverse Events (participants affected / at risk) | 81/82 | 80/81 | 82/82 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=82) | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (N=81) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (N=82) | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week (N=78)
RASH (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 3 | 1 | 1
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 2
DISORIENTATION (Psychiatric disorders) | 0 | 0 | 0 | 1
EMOTIONAL DISTRESS (Psychiatric disorders) | 0 | 0 | 1 | 0
PARANOIA (Psychiatric disorders) | 1 | 0 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 1
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA HERPES VIRAL (Infections and infestations) | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 1 | 1 | 1
SPEECH DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
ASTHENIA (General disorders) | 0 | 1 | 0 | 0
CATHETER RELATED COMPLICATION (General disorders) | 0 | 0 | 1 | 0
CHILLS (General disorders) | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TESTICULAR SWELLING (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 0
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 1
SPLENECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=82) | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (N=81) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (N=82) | Telaprevir 12 Week+Peg-IFN-alfa-2a 12 Week (N=78)
ASTHENIA (General disorders) | 26 | 37 | 43 | 30
INFLUENZA LIKE ILLNESS (General disorders) | 43 | 32 | 32 | 28
Fatigue (General disorders) | 30 | 21 | 23 | 26
PYREXIA (General disorders) | 19 | 14 | 15 | 15
IRRITABILITY (General disorders) | 11 | 7 | 7 | 8
CHILLS (General disorders) | 10 | 1 | 6 | 5
INJECTION SITE ERYTHEMA (General disorders) | 3 | 2 | 4 | 6
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 2 | 3 | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 29 | 41 | 52 | 46
DRY SKIN (Skin and subcutaneous tissue disorders) | 29 | 21 | 21 | 22
RASH (Skin and subcutaneous tissue disorders) | 22 | 27 | 23 | 21
ALOPECIA (Skin and subcutaneous tissue disorders) | 17 | 15 | 3 | 11
ECZEMA (Skin and subcutaneous tissue disorders) | 5 | 10 | 13 | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 7 | 5 | 7
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 4 | 5 | 4 | 6
NAUSEA (Gastrointestinal disorders) | 33 | 39 | 39 | 24
DIARRHOEA (Gastrointestinal disorders) | 23 | 20 | 26 | 20
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 8 | 8 | 7
VOMITING (Gastrointestinal disorders) | 12 | 10 | 5 | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 | 8 | 6 | 5
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 9 | 10 | 5
DRY MOUTH (Gastrointestinal disorders) | 4 | 1 | 9 | 6
ANAL PRURITUS (Gastrointestinal disorders) | 0 | 6 | 9 | 4
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 2 | 4 | 9 | 3
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 5 | 2
HEADACHE (Nervous system disorders) | 37 | 36 | 32 | 37
DYSGEUSIA (Nervous system disorders) | 3 | 5 | 11 | 4
DIZZINESS (Nervous system disorders) | 8 | 5 | 6 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 2 | 5 | 4 | 7
LETHARGY (Nervous system disorders) | 4 | 1 | 2 | 4
INSOMNIA (Psychiatric disorders) | 32 | 23 | 28 | 11
DEPRESSION (Psychiatric disorders) | 19 | 16 | 18 | 17
ANXIETY (Psychiatric disorders) | 3 | 4 | 5 | 5
NERVOUSNESS (Psychiatric disorders) | 4 | 1 | 6 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 17 | 11 | 12 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 | 8 | 8 | 20
INFLUENZA (Infections and infestations) | 6 | 9 | 2 | 8
NASOPHARYNGITIS (Infections and infestations) | 8 | 5 | 5 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 16 | 5 | 9 | 16
ANOREXIA (Metabolism and nutrition disorders) | 2 | 4 | 5 | 1
DRY EYE (Eye disorders) | 4 | 5 | 5 | 2
WEIGHT DECREASED (Investigations) | 6 | 5 | 2 | 4
VERTIGO (Ear and labyrinth disorders) | 11 | 6 | 7 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 18 | 21 | 11
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 15 | 14 | 8
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 7 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 4 | 4 | 10
BRONCHITIS (Infections and infestations) | 1 | 1 | 1 | 4
ANAEMIA (Blood and lymphatic system disorders) | 14 | 22 | 15 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 14 | 3 | 6 | 2
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days